CLINICAL TRIAL: NCT01463709
Title: Development of a Nanosecond Pulsed Electric Field System to Treat Skin Cancer
Acronym: NPEF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-049
Record Dates: First submitted 2011-10-26; First posted 2011-11-02 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Basal Cell Carcinomas
Keywords: basal cell carcinoma; Basal Cell Nevus Syndrome; Electric Field; Nanosecond pulse
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanopulse (Experimental): Administer nano pulse to lesion for varying time intervals.
  Interventions: Device: PulseCure pulse generator and Derm-pulse electrode

INTERVENTIONS:
Device: PulseCure pulse generator and Derm-pulse electrode — PulseCure 100 ns pulse generator: generates 30 kV/cm electric pulses 100 ns long to trigger apoptosis in cells between the electrodes.
  NanoBlate: Delivery device to treat 5 mm wide skin lesions with 100 ns pulses from PulseCure
  Other Names: BioElectroMed

SUMMARY:
Human Basal Cell Carcinomas (BCCs) can be ablated by treating them with nanosecond pulsed electric fields (nsPEF)

DETAILED DESCRIPTION:
The purpose of this study is to determine if low energy, non-thermal, 100 ns pulses can ablate BCCs. The investigators consider this a non-significant risk study because our PulseCure system only applies 0.4 watts to the skin compared to the 40 watts applied by the currently used electrosurgical unit to remove skin lesions, the Hyfrecator. Since the PulseCure applies 1/100 of the energy and does not even heat the skin significantly, it represents a non-significant risk to the patient. Our study will provide the first data on the response of BCCs to these 100 ns pulses. The investigators will first treat three BCCs on BCNS patients with different pulse numbers to determine the pulse number needed to ablate. Once the investigators have the optimal pulse number, the investigators will use it to treat 20 normal patients with sporadic BCCs on their trunks. This should provide sufficient data to conclude whether or not nsPEF can ablate BCCs on normal individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Study subjects must have had diagnosed at least one BCCon their trunk
2. The subject is from 18-75 years of age, inclusive.
3. The subject must sign and date all informed consent statements.

Exclusion Criteria:

1. The subject is exhibiting signs of a bacterial or viral infection, including fever.
2. The subject is unwilling to allow a biopsy of a malignant lesion for histological analysis.
3. The subject has a pace maker or other electronic device implanted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the safety of PulseCure pulse generator and NanoBlate electrode and identify the optimal pulse number for treating basal cell carcinomas. | One year
  1. Conduct a non-significant risk feasibility clinical trial treating BCCs on the trunk of up to 9 Basal Cell Nevus Syndrome patients with BioElectroMed's PulseCure pulse generator and Derm-Pulse electrode to both demonstrate the safety of nsPEF therapy and identify the optimal pulse number for ablating BCCs.

SECONDARY OUTCOMES:
Determine the efficacy of the PulseCure pulse generator using the optimal pulse number. | one year
  2. Conduct a non-significant risk Pilot Clinical Trial treating BCCs on the trunk of 20 patients with sporadic BCCs using the optimal pulse number determined from the feasibility trial to assess the efficacy of this technique.

CONTACTS AND LOCATIONS:
Overall Officials: Ervin E Epstein, MD, Principal Investigator — Children's Hospital Research Institute
Locations (1):
- Children's Hospital Research Center Oakland, Oakland, California, United States